CLINICAL TRIAL: NCT06001996
Title: The Effects of Pericapsular Nerve Group (PENG) Block and Fascia Iliaca Plane Block on Preoperative and Postoperative Analgesia Before Spinal Anaesthesia in Patients Undergoing Hip Fracture Surgery
Brief Title: Comparison of Intraoperative- Postoperative Effects of Pericapsular Nerve Block and Fascia Iliaca Block in Hip Fracture
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 12.09.2022/265
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pericapsular nerve group (PENG) block: Group 1:Pericapsular nerve group (PENG) block: Using an in-plane approach with ultrasonographic imaging, the block needle reaches the fascial plane between the psoas muscle and the upper pubic ramus, and patients injected with local anesthetic solution.
  * After the patients were sedated with intravenous 1 mg midazolam and 50 mcg fentanyl in the preoperative preparation room, 15 ml of 0.375% bupivacaine was administered to the fractured hip side under ultrasound guidance.
  * After the block application, the patient will be taken to the operating room and standard spinale anaesthesia will be applied.
  * Each patient will receive 15 ml of 0.375% bupivacaine 0.375% on the side of the broken hip only one time approximately 15-20 minutes before the operation.
  * Plane block applications will be applied only once in the preoperative period
  * Plane block applications will be performed by anaesthesiologists with at least 5 years of experience
  Interventions: Procedure: Pericapsular nerve group (PENG) block
- Suprainguinal fascia iliaca plane block: Group 2: Suprainguinal fascia iliaca plane block: Patients in whom the needle entered in plane from the caudal end of the ultrasound probe passes through the musculus iliacus and fascia iliaca and local anesthetic solution has been injected immediately under the fascia.
  After the patients were sedated with intravenous 1 mg midazolam and 50 mcg fentanyl in the preoperative preparation room, 15 ml of 0.375% bupivacaine was administered to the fractured hip side under ultrasound guidance. After the block application, the patient will be taken to the operating room and standard spinale anaesthesia will be applied.
  Each patient will receive 15 ml of 0.375% bupivacaine 0.375% on the side of the broken hip only one time approximately 15-20 minutes before the operation.
  * Plane block applications will be applied only once in the preoperative period
  * plane block applications will be performed by anaesthesiologists with at least 5 years of experience
  Interventions: Procedure: Suprainguinal fascia iliaca plane block

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block — Pericapsular nerve group (PENG) block: Using an in-plane approach with ultrasonographic imaging, the block needle reaches the fascial plane between the psoas muscle and the superior pubic ramus and local anaesthetic solution is injected.
  Groups: Pericapsular nerve group (PENG) block
Procedure: Suprainguinal fascia iliaca plane block — Suprainguinal fascia iliaca plane block: The needle entering in plane from the caudal end of the ultrasound probe passes through the m. sartorius and into the musculus iliacus and fascia iliaca reaches. The fascia iliaca is passed with the needle and local anaesthetic solution is injected immediately under the fascia.
  Groups: Suprainguinal fascia iliaca plane block

SUMMARY:
The aim of this study is to apply pericapsular nerve group (PENG) block or fascia iliaca plan block using ultrasonography to patients who will undergo hip fracture surgery, while giving sitting position before spinal anaesthesia and to reduce postoperative pain complaints.

Thanks to these blocks, it is aimed to reduce pain complaints and the need for morphine-derived painkillers before and after surgery.

DETAILED DESCRIPTION:
Group 1:Pericapsular nerve group (PENG) block: Using an in-plane approach with ultrasonographic imaging, the block needle reaches the fascial plane between the psoas muscle and the superior pubic ramus and local anaesthetic solution is injected.

* Each patient will receive 15 ml of 0.375% bupivacaine on the side of the broken hip only one time approximately 15-20 minutes before the operation.
* After the patients were sedated with intravenous 1 mg midazolam and 50 mcg fentanyl in the preoperative preparation room, 15 ml of 0.375% bupivacaine was administered to the fractured hip side under ultrasound guidance. After the block application, the patient will be taken to the operating room and standard spinale anaesthesia will be applied.
* plane block applications will be performed by anaesthesiologists with at least 5 years of experience
* Postoperative evaluations of patients will be performed face to face.
* Plane block applications will be applied only once in the preoperative period.
* Patients will be routinely administered 1 g paracetamol intravenously at 8 hour intervals in the postoperative period. 100 mg tramadol intravenously will be administered if their pain is above Numerical Rating Scale (NRS) 4 despite this.
* This study was followed up in the orthopaedic service
* Patients will be monitored for pain and side effects at the postanesthetic care unit , 1st hour, 2nd hour, 4th hour, 8th hour and 24th hour in the postoperative period.
* The extent to which plan blocks facilitate the positioning of the patient for spinal anaesthesia in the intraoperative period will be monitored. In addition, the effects on intraoperative and postoperative opioid consumption and patient satisfaction will be observed.
* Data on the observed parameters will be obtained from face-to-face questionnaires or anesthesia and nurse observation forms.

Group 2: Suprainguinal fascia iliaca plane block: The needle entering in plane from the caudal end of the ultrasound probe passes through the m. sartorius and into the musculus iliacus and fascia iliaca reaches. The fascia iliaca is passed with the needle and local anaesthetic solution is injected immediately under the fascia.

* Each patient will receive 15 ml of 0.375% bupivacaine on the side of the broken hip only one time approximately 15-20 minutes before the operation.
* After the patients were sedated with intravenous 1 mg midazolam and 50 mcg fentanyl in the preoperative preparation room, 15 ml of 0.375% bupivacaine was administered to the fractured hip side under ultrasound guidance. After the block application, the patient will be taken to the operating room and standard spinale anaesthesia will be applied.
* plane block applications will be performed by anaesthesiologists with at least 5 years of experience
* Postoperative evaluations of patients will be performed face to face.
* Plane block applications will be applied only once in the preoperative period.
* Patients will be routinely administered 1 g paracetamol intravenously at 8 hour intervals in the postoperative period. 100 mg tramadol intravenously will be administered if their pain is above Numerical Rating Scale (NRS) 4 despite this.
* This study was followed up in the orthopaedic service.
* Patients will be monitored for pain and side effects at the postanesthetic care unit , 1st hour, 2nd hour, 4th hour, 8th hour and 24th hour in the postoperative period.
* The extent to which plan blocks facilitate the positioning of the patient for spinal anaesthesia in the intraoperative period will be monitored. In addition, the effects on intraoperative and postoperative opioid consumption and patient satisfaction will be observed.
* Data on the observed parameters will be obtained from face-to-face questionnaires or anesthesia and nurse observation forms.
* Statistical methods / analysis: G-Power version 3.1.9.4 (University Kiel, Germany) program was used to calculate the sample size. The two-tailed alpha error was taken as 0.05, power as 0.80 and effect size as 0.8, and based on a previous study the allocation ratio was accepted as N2/N1:1. The minimum number of patients to be included in the study was calculated as 52.

SPSS 16.0 for Windows (SPSS Inc., Chicago, USA) was used for other statistical analyses. Statistical data were expressed as mean and standard deviation, while categorical data were expressed as frequency and percentage. Comparison of categorical data in the groups was done with Chi-square, the results were given as %n. Shapiro-Wilk tests were used to determine if the numerical data fit the normal distribution. While the data fitting the normal distribution were evaluated with the Student's t-test. Mann- Whitney U tests were used to compare the data differ from the normal distribution. p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years of age,
* American Society of Anesthesiologists (ASA) Classification I-III,
* scheduled for hip fracture surgery under spinal anaesthesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Classification >III
* known allergy to local anaesthetics
* presence of preoperative chronic pain
* presence of coagulopathy
* those who are unable to give written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip fracture
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Assessment of pain level | 1: measured in neutral position before the block. 2: measured with 15 degrees elevation of the affected limb before the block.3: Measured in spinal positioning. 4: Measured between 0-2 hours postoperatively. 5: Measured between 2-8 hours postoperatively
  Assessment of pain level with the Numerical Rating Scale (NRS) :
  The 11-point numerical scale ranges from '0' representing one pain end (e.g. "no pain") to '10' representing the other pain end (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Evaluation of ease of positioning | Procedure (at the stage of introduction of spinal anaesthesia)
  It was determined by means of a scale scored from 0-3 (0=no positioning, 1=standing in abnormal posture due to pain and needing support for positioning 2=mild discomfort but no need for support for positioning 3=able to position on their own without pain).

SECONDARY OUTCOMES:
Agitation assessment | During positioning for spinal anaesthesia procedure
  Agitation assessment with Richmond Agitation Sedation Scale (RASS) is a 10-point scale ranging from -5 to +4.Levels -1 to -5 denote 5 levels of sedation, starting with "awakens to voice" and ending with "unarousable." Levels +1 to +4 describe increasing levels of agitation. The lowest level of agitation starts with apprehension and anxiety, and peaks at combative and violent. RASS level 0 is "alert and calm.
mean blood pressure | Intraoperative (1- Baseline 2- During spinal block 3- 5th minutes after spinal block 4- Every 10 minutes during the operation 5- Skin closure)
  Mean blood pressure assessed using automatic sphygmomanometer over a 60 second interval
Heart rate | Intraoperative (1- Baseline 2- During spinal block 3- 5th minutes after spinal block 4- Every 10 minutes during the operation 5- Skin closure)
  The number of heart beats per minute obtained by electrocardiographic monitoring
Tramadol consumption after surgery | 24 hours postoperatively
  Total amount of tramadol consumed within 24 hours after surgery
Time of first analgesia use | up to 24 hours (Duration of the first analgesic requirement after surgery (in hours))
  Duration of the first analgesic requirement after surgery (in hours)
Limb range of motion | 1- Postoperative 4th hours , 2- Postoperative 8th hours
  Limb range of motion assessed using goniometer
Patient satisfaction score | Second postoperative day
  Patients' satisfaction with the quality of pain management will be assessed on the second postoperative day using the following scale: 1 = very unsatisfied; 2 = quite unsatisfied; 3 = moderate; 4 = quite satisfactory; 5 = very satisfactory.
Number of Participants with Side effects | within 24 hours postoperatively
  Number of Participants with side effects such as neurological deficit, oedema, haematoma, nausea and vomiting will be evaluated by physical examination, patient anamnesis and nurse follow-up forms

CONTACTS AND LOCATIONS:
Overall Officials: Cem K. Kaçar, Assoc.Prof, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi YS, Park KK, Lee B, Nam WS, Kim DH. Pericapsular Nerve Group (PENG) Block versus Supra-Inguinal Fascia Iliaca Compartment Block for Total Hip Arthroplasty: A Randomized Clinical Trial. J Pers Med. 2022 Mar 6;12(3):408. doi: 10.3390/jpm12030408. PMID 35330408